CLINICAL TRIAL: NCT06163898
Title: A Phase 1b/2a, Multicenter, Open-label Study to Determine the Recommended Dose and Schedule, and Evaluate the Safety and Preliminary Efficacy of Alnuctamab in Combination With Mezigdomide in Participants With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study to Evaluate Alnuctamab in Combination With Mezigdomide in Participants With Relapsed and/or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA058-002; 2023-504367-16-00 (Other: EU CTR); U1111-1283-8970 (Other: WHO)
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A (Experimental)
  Interventions: Drug: Alnuctamab; Drug: Mezigdomide; Drug: Dexamethasone
- Arm B1 (Experimental)
  Interventions: Drug: Alnuctamab; Drug: Mezigdomide; Drug: Dexamethasone
- Arm B2 (Experimental)
  Interventions: Drug: Alnuctamab; Drug: Mezigdomide; Drug: Dexamethasone
- Arm C1 (Experimental)
  Interventions: Drug: Alnuctamab; Drug: Mezigdomide; Drug: Dexamethasone
- Arm C2 (Experimental)
  Interventions: Drug: Alnuctamab

INTERVENTIONS:
Drug: Alnuctamab — Specified dose on specified days
  Other Names: BMS-986349; CC-93269; EM901
Drug: Mezigdomide — Specified dose on specified days
  Other Names: BMS-986348; CC-92480
  Arms: Arm B1; Arm B2; Arm C1; Part A
Drug: Dexamethasone — Specified dose on specified days
  Arms: Arm B1; Arm B2; Arm C1; Part A

SUMMARY:
The purpose of this study is to determine the recommended dose and schedule, and evaluate the safety and preliminary efficacy of alnuctamab in combination with mezigdomide in participants with relapsed and/or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

Participant has a history of RRMM, and must:

* Part A: Have previously received ≥ 3 prior lines of anti-myeloma therapy.
* Part B and Part C: Have received 1 to 3 prior lines of anti-myeloma therapy.

Exclusion Criteria:

• Must not have previously received alnuctamab or mezigdomide.

Note: Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up until 28 days after the last participant discontinues mezigdomide or 80 days after the last participant discontinues alnuctamab, whichever is longer (up to approximately 5 years)
Number of participants with serious AEs (SAEs) | Up until 28 days after the last participant discontinues mezigdomide or 80 days after the last participant discontinues alnuctamab, whichever is longer (up to approximately 5 years)
Number of participants with AEs leading to discontinuation | Up until 28 days after the last participant discontinues mezigdomide or 80 days after the last participant discontinues alnuctamab, whichever is longer (up to approximately 5 years)
Number of deaths | Up until 28 days after the last participant discontinues mezigdomide or 80 days after the last participant discontinues alnuctamab, whichever is longer (up to approximately 5 years)
Number of participants with Dose-limiting toxicities (DLTs) | Up until 28 days after the last participant discontinues mezigdomide or 80 days after the last participant discontinues alnuctamab, whichever is longer (up to approximately 5 years)
Overall Response Rate (ORR) | From first participant enrollment until the last participant is no longer evaluable for response, or has progressed or the last survival follow-up (Up to approximately 5 years)
  Phase 2 only

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | From first participant enrollment until the last participant is no longer evaluable for response, or has progressed or the last survival follow-up (Up to approximately 5 years)
Very Good Partial Response Rate (VGPRR) | From first participant enrollment until the last participant is no longer evaluable for response, or has progressed or the last survival follow-up (Up to approximately 5 years)
Progression-free Survival (PFS) | From first participant enrollment until the last participant is no longer evaluable for response, or has progressed or the last survival follow-up (Up to approximately 5 years)
Time-to-Response (TTR) | From first participant enrollment until the last participant is no longer evaluable for response, or has progressed or the last survival follow-up (Up to approximately 5 years)
Duration of Response (DOR) | From first participant enrollment until the last participant is no longer evaluable for response, or has progressed or the last survival follow-up (Up to approximately 5 years)
Overall Survival (OS) | From first participant enrollment until the last participant is no longer evaluable for response, or has progressed or the last survival follow-up (Up to approximately 5 years)
ORR | From first participant enrollment until the last participant is no longer evaluable for response, or has progressed or the last survival follow-up (Up to approximately 5 years)
  Phase 1 only

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (3):
  - Local Institution - 0033, Birmingham, Alabama
  - Local Institution - 0035, New Haven, Connecticut
  - Local Institution - 0018, New York, New York
- Israel (3):
  - Local Institution - 0021, Petah Tikva, Central District
  - Local Institution - 0030, Ramat Gan, Central District
  - Local Institution - 0020, Jerusalem

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html